CLINICAL TRIAL: NCT04643938
Title: Preimplantation Genetic Testing for Aneuploidy in Screening of Embryos in the Treatment of Unexplained Recurrent Miscarriage: a Single-center, Prospective Clinical Analysis Based on aCGH Technology
Brief Title: PGT-A in Screening of Embryos in the Treatment of Unexplained Recurrent Miscarriage
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Wang Haiyan, Professor, Peking University Third Hospital
Other Study IDs: 2019SZ-076
Record Dates: First submitted 2020-11-03; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Recurrent Early Pregnancy Loss
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Two spontaneous abortions: No intervention
- three spontaneous abortions: No intervention
- Four or more spontaneous abortions: No intervention

SUMMARY:
uRM patients selected PGT-A from 2012 to 2016 were included in this study. Their clinical outcomes were prospectively observed and analyzed to explore the factor influenced the outcomes.

DETAILED DESCRIPTION:
This prospective observational study enrolled all women with uRM who underwent array-comparative genomic hybridization (array-CGH) for PGT-A in the Reproductive Medicine Center of Peking University Third Hospital from 2012 to 2016. If a couple underwent multiple stimulation cycles during the research period, only the first cycle was included. All patients underwent adequate clinical and genetic consultations before undergoing PGT-A, and all voluntarily chose PGT-A after fully understanding its risks and benefits. All patients signed the informed consent document of PGT-A. All included stimulation cycles involved intracytoplasmic sperm injection insemination. After successfully fertilized embryos formed blastocysts on Day 5-7, trophoblasts were biopsied to determine embryonic karyotypes. The blastocysts with normal/balanced test results were cryopreserved, whereas abnormal blastocysts were discarded after notifying the patients. All normal blastocysts from a patient were thawed and transferred singly, and the outcomes of all subsequent frozen-thawed embryo transfer cycles were followed-up until January 2020.

Clinical outcomes included the blastocyst formation rate, the proportion of blastocysts with normal karyotypes, and the clinical pregnancy, live birth, and cumulative live birth rates. The factors that affected these clinical outcomes were analyzed to predict outcomes and guide treatment in women with uRM.

ELIGIBILITY:
Inclusion Criteria:

women with uRM who underwent array-comparative genomic hybridization (array-CGH) for PGT-A in the Reproductive Medicine Center of Peking University Third Hospital from 2012 to 2016.Only the first cycle was included. All patients underwent adequate clinical and genetic consultations before undergoing PGT-A, and all voluntarily chose PGT-A after fully understanding its risks and benefits. All patients signed the informed consent document of PGT-A.

Exclusion Criteria:

Couples with parental chromosomal abnormalities were excluded, as were women with anatomical abnormalities of the uterus, autoimmune diseases, and endocrine abnormalities.

Ages: 20 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Both biological and social sexes are female
Study Population: women with uRM who underwent array-comparative genomic hybridization (array-CGH) for PGT-A in the Reproductive Medicine Center of Peking University Third Hospital from 2012 to 2016
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Baseline characteristics | January 2012 to December 2016
  Age
Baseline characteristics | January 2012 to December 2016
  basal sex hormone
Baseline characteristics | January 2012 to December 2016
  the number of abortion
laboratory outcomes of patients | January 2012 to December 2016
  Oocyte count
laboratory outcomes of patients | January 2012 to December 2016
  Number of blastocysts
clinical outcoms | January 2012 to January 2020
  normal karyotype blastocyst rate
clinical outcoms | January 2012 to January 2020
  live birth rate
clinical outcoms | January 2012 to January 2020
  Cumulative pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Wang, M.D., Principal Investigator — Center of Reproductive Medicine, Peking University Third Hospital
Locations (1):
- Center of Reproductive Medicine, Peking University Third Hospital, Beijing, Haidian, China

IPD SHARING:
Plan to Share IPD: No